CLINICAL TRIAL: NCT05402852
Title: Effectiveness and Safety of EuBone® Capsules for Bone Health in Postmenopausal Women：A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effectiveness and Safety of EuBone® Capsules for Bone Health in Postmenopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Qianfoshan Hospital (Other); Chenland Nutritionals lnc. (Unknown); Jinan Hetai Pharmaceutical Technology Co., LTD (Unknown)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-PD-2021-08
Record Dates: First submitted 2022-05-22; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: Subjects were randomly assigned to the EuBone® capsule treatment group or placebo control group in a 2:1 ratio.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug：EuBone® capsule (Experimental): Subjects are given EuBone® capsules, 4 capsules ×500mg/capsule per day for 360 days.
  Interventions: Drug: EuBone ® capsule
- control：placebo (Placebo Comparator): Subjects are given placebo capsules, 4 capsules ×500mg/capsule per day for 360 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EuBone ® capsule — Subjects are given EuBone® capsules, 4 capsules ×500mg/capsule per day for 360 days.
  Arms: Drug：EuBone® capsule
Drug: placebo — Subjects are given placebo capsules, 4 capsules ×500mg/capsule per day for 360 days.
  Arms: control：placebo

SUMMARY:
EuBone is prepared by mixing eucommia ulmoides extract, fructus ulmoides extract and dodder extract in proportion. The aim of this study is to evaluate the effectiveness and safety of EuBone® capsules in slowing bone loss, preventing bone loss, and improving quality of life compared with placebo in Postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign written informed consent and comply with the requirements and restrictions of the test;
* Female subjects；Age: 45-75 years (including boundary values)；Menopause ≥12 months；Not receiving hormone replacement therapy;
* Meet the bone reduction criteria: -2.5<T value<-1.0；
* OSTA index < -1, OSTA index = [body weight (kg) - age (years)] ×0.2;
* Have the ability of independent activities。

Exclusion Criteria:

* Patients with abnormalities in lumbar vertebra, hip bone and femoral neck cannot be measured by BMD;
* Patients with osteoporosis, BMD T-score of the whole hip, femoral neck or lumbar spine ≤-2.5;
* Have the following diseases known to affect calcium or bone metabolism: various metabolic bone diseases, such as osteogenesis imperfecta, osteomalacia; Paget's disease of bone; Cushing's syndrome; Hyperprolactitinemia; Hypopituitarism; Acromegaly; Rheumatoid arthritis; History of hyperparathyroidism or hypoparathyroidism;
* Patients who are suffering from or have suffered from osteomyelitis or osteonecrosis of the jaw, or who plan to undergo invasive dental surgery or jaw surgery during the trial, or who have unhealed dental or oral surgery wounds;
* Fractures in the past 6 months;
* People with allergic constitution, or known allergy to the test drug ingredients, or a history of allergy to any drug, food or pollen;
* Randomized prior or plan to use drugs that may affect bone turnover during the study period, including, but not limited to, the following: Used denumab , bisphosphonate or fluoride in the last 12 months, used Contraceptive pills containing estrogen, hormone replacement therapy (e.g., Tibolone, estrogen and selective estrogen receptor modulators, etc.), aromatase inhibitors, calcitonin, strontium salt, parathyroid hormone (or derivative), vitamin D supplements (> 1000 IU/ day), anabolic steroids, systemic glucocorticoids, calcitriol or analogues, diuretics, anticonvulsants in the last 6 months; Use inhaled or topical glucocorticoid drugs within 2 weeks;
* Had significant changes in physical activity within 6 months prior to randomization, or had been engaged in vigorous physical exercise, or planned to participate in vigorous physical exercise during the trial;
* Hepatitis B virus surface antigen (HBsAg), anti-hepatitis C virus antibody (HCV-AB), anti-HIV and anti-treponema pallidum antibody (TP-AB) are positive;
* Hypocalcemia or hypercalcemia, or serum albumin-corrected serum calcium levels not within the laboratory normal range;
* After inquiry, the average daily smoking quantity within 3 months prior to randomization ≥5, or can not stop smoking during the trial period;
* Binge drinking or drinking more than 28 units of alcohol per week (1 unit =350ml beer or 45ml spirits or 150ml wine) within 3 months prior to randomization;
* Have a history of drug abuse or drug abuse;
* Complete blood donation, component blood donation, or massive bleeding (>400 ml) within 3 months prior to randomization;
* Participants in interventional clinical trials of other drugs or devices within 3 months prior to randomization;
* Suffering from other important primary diseases (such as diseases of the nervous system, cardiovascular system, urinary system, digestive system, respiratory system or metabolic endocrine system) that are not considered suitable for admission, or for other reasons that are not considered suitable for admission;
* Other factors that the researcher considers unsuitable for inclusion.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The response rate of Quality of life score from baseline | on day 360 after administration
  To evaluate the improvement rate of the Quality of life score from baseline improvement rate
The change of lumbar vertebra bone density | on day 360 after administration
  To evaluate the change of lumbar vertebra bone density from baseline
The incidence rate of adverse events | Through study completion, an average of 360 days
  To evaluate the incidence rate of adverse events

SECONDARY OUTCOMES:
The response rate of quality of life score | at 30, 90 and 180 days after administration
  To evaluate the improvement rate of quality of life score from baseline
The change of bone mineral density (BMD) at the total hip joint and femoral neck of the subject | at 180 and 360 days after continuous administration of EuBone® capsule
  To evaluate the change of bone mineral density (BMD) at the total hip joint and femoral neck of the subject after continuous administration of EuBone® capsule compared from baseline
The change of bone mineral density of lumbar vertebra (L1~L4) | at 180 after continuous administration of EuBone® capsule
  To evaluate the change of bone mineral density of lumbar vertebra (L1~L4) after continuous administration of EuBone® capsule
The change of serum n-terminal propeptide (S-PINP) and carboxy-terminal cross-linked peptide of type I procollagen (S-CTX) from baseline | at 30, 90, 180 and 360 days after administration
  To evaluate the change of serum n-terminal propeptide (S-PINP) and carboxy-terminal cross-linked peptide of type I procollagen (S-CTX) in EuBone® capsule from baseline
The change of parathyroid hormone (PTH), calcitonin (CT) and estrogen levels | at 30, 90, 180 and 360 days after administration
  To evaluate the changes of parathyroid hormone (PTH), calcitonin (CT) and estrogen levels after continuous treatment with EuBone® capsule from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Ji'nan, Shandong, China